CLINICAL TRIAL: NCT06885918
Title: ALS Translational Research Program
Brief Title: ALS Research Collaborative
Acronym: ARC
Status: Recruiting | Type: Observational
Sponsor: ALS Therapy Development Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ALSTDI0103
Record Dates: First submitted 2025-02-27; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS (Amyotrophic Lateral Sclerosis); ALS With Frontotemporal Dementia (ALS/FTD); Motor Neuron Disease; Motor Neuron Disease, Amyotrophic Lateral Sclerosis
Keywords: ARC; ALS Research Collaborative; ALS TDI; ALS Therapy Develeopment Institute
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; AIDS-Related Complex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Fibroblasts, Serum, Plasma, Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Person living with ALS/MND: An adult over the age of 18, that has received a diagnosis of ALS or other Motor Neuron Disease from a practicing physician.
- Asymptomatic gene carrier: An adult over the age of 18 who does not have symptoms of ALS and carries a mutation known to be associated with ALS
- Healthy Volunteer: An adult over the age of 18 who does not have any biological connection to ALS or other Motor Neuron Disease, and no significant health problems.

SUMMARY:
The goal of this natural history study is to learn more about the biological and clinical aspects of amyotrophic lateral sclerosis (ALS). This study's findings will help with drug discovery, biomarker discovery, and outcome measure validation. Adults living with ALS, other motor neuron diseases (MND), a known mutation related to ALS and healthy volunteers contribute prospective and retrospective data to this study remotely. The study is sponsored and conducted by the ALS Therapy Development Institute.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Can communicate in written English
* Has a diagnosis of ALS/MND or is a known carrier of an ALS associated mutation

Exclusion Criteria:

* Significant cognitive impairment that would prevent individual completion and understanding of the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants can be located anywhere but require internet access.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-09-12 (Actual); Primary Completion 2035-01-31 (Estimated); Study Completion 2035-01-31 (Estimated)

PRIMARY OUTCOMES:
ALS Functional Rating Scale - Revised (ALSFRS-R) | Monthly, through study completion, an average of 1 year
  A questionnaire completed by the participant that assesses 12 daily functions of living on a 0 (severe symptoms) to 4 (minimal to no symptoms) integer scale.

SECONDARY OUTCOMES:
Machine-Learning Based Speech Scoring | Monthly, through study completion, an average of 1 year
  Participants submit a scripted voice recording of 5 different, short phrases that are then scored by a machine-learning based algorithm that assess dysarthria on a non-integer scale of 0 (fully impaired) to 4 (normal speech)
Limb-based Accelerometry | monthly, through study completion, an average of 6 months
  Participants wear four, ActiGraph devices on each limb. Passive and active (video-directed) wear time data is collected over one week. The devices measure acceleration and represent the strength of each limb during movement. Outputs include activity counts and raw acceleration data.
Medications, Supplements, and Clinical Trial Participation Surveys | quarterly, through study completion, an average of 1 year
  Participants complete questionnaires describing usage information about medications and supplements they have taken and are currently taking, as well as clinical trial participation.
Social and Environmental Surveys | One-time or quarterly at months 1, 4, 7, 10
  Participants complete questionnaires about their familial, educational, and geographical background, as well as lifestyle habits and past medical conditions and injuries. These are non-current factors that may have an affect on current health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando G Vieira, M.D., Principal Investigator — ALS Therapy Development Institute
Locations (1):
- ALS Therapy Development Institute, Watertown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Straczkiewicz M, Burke KM, Calcagno N, Premasiri A, Vieira FG, Onnela JP, Berry JD. Free-living monitoring of ALS progression in upper limbs using wearable accelerometers. J Neuroeng Rehabil. 2024 Dec 21;21(1):223. doi: 10.1186/s12984-024-01514-7. PMID 39707523
- [Background] Gupta AS, Patel S, Premasiri A, Vieira F. At-home wearables and machine learning sensitively capture disease progression in amyotrophic lateral sclerosis. Nat Commun. 2023 Aug 21;14(1):5080. doi: 10.1038/s41467-023-40917-3. PMID 37604821
- [Background] Vieira FG, Venugopalan S, Premasiri AS, McNally M, Jansen A, McCloskey K, Brenner MP, Perrin S. A machine-learning based objective measure for ALS disease severity. NPJ Digit Med. 2022 Apr 8;5(1):45. doi: 10.1038/s41746-022-00588-8. PMID 35396385
- See also: ARC Sign Up Page — https://arc.als.net/
- See also: ARC Data Commons Inquiry Page - for researcher access to ARC data — https://www.als.net/arc/data-commons/